CLINICAL TRIAL: NCT06323538
Title: Cohort Study on Plant-based Diets (COPLANT Study)
Acronym: COPLANT
Status: Recruiting | Type: Observational
Sponsor: German Federal Institute for Risk Assessment (Other)
Collaborators: Max Rubner-Institut (Unknown); University of Bonn (Other); Research Institute for Plant-Based Nutrition (Unknown); University of Jena (Other); University of Regensburg (Other); Heidelberg University (Other); University of Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: 01
Record Dates: First submitted 2024-03-01; First posted 2024-03-21 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Dietary Exposure; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Bone Loss; Sustainability; Exposure; Obesity; Vitamin Deficiency; Mineral Deficiency
Keywords: vegan; vegetarian; pescetarian; omnivor; multicenter cohort; biomarker; vitamins; minerals; bone health; cardiovascular risk; body composition; inflammation; contaminants; diabetes type 2; thyroid gland health; microbiota; metabolomics; adults; children; pregnancy; breast feeding time; mental health; sustainability
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Bone Diseases, Metabolic; Obesity; Avitaminosis; Inflammation; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fasting blood samples, 24h urine, stool samples, saliva, breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- vegans: vegan diet: no products of animal origin
- vegetarians: vegetarian diet: no meat and fish, but dairy products and eggs
- pescetarians: pescetarian diet: no meat, but fish
- mixed diet: mixed diet: plant-based foods and animal-based foods

SUMMARY:
The Cohort on Plant-based Diets (COPLANT) study is a multi-centre cohort study that starts baseline recruitment from 2024 to 2027 with approximately 6,000 participants in Germany and Austria. The COPLANT study focuses on vegan (no animal products), vegetarian (no meat and fish, but dairy products and eggs), pescetarian (no meat, but fish) and omnivorous (mixed diet including all possible animal products) diets. The aim of the COPLANT study is to gain new insights on health benefits and risks as well as social, ecological and economic effects of different plant-based diets in comparison to a mixed diet. In addition to a detailed dietary survey using an app adapted to the needs of this study, the baseline examination includes measurements of body composition, bone health, cardiovascular risk factors, diabetes risk, contaminants and lifestyle. For the basic laboratory program, fasting blood, 24-hour urine collection and a stool sample are taken from all study participants. Furthermore, specific aspects of dietary behavior, physical activity and other lifestyle factors are collected via questionnaires. Follow-up studies are planned at intervals of 5, 10 and 20 years after the baseline visit.

DETAILED DESCRIPTION:
The multicenter Cohort on Plant-based diets (COPLANT) study, aims to investigate the health benefits as well as short-term and long-term risks of different plant-based diets (vegan: no animal products, vegetarian: no meat and fish, but dairy products and eggs, pescetarian: no meat, but fish) compared to a mixed diet among 6,000 participants aged 18 to 69 years across German speaking countries. Currently the impact of different diets not only on health effects, but also on social, ecological and economic factors is becoming increasingly evident in areas of social justice, climate change and animal welfare. For this reason, a sustainability analysis (social, ecological and economic effects) together with findings on health effects will be included in the COPLANT study. As plant-based diets, especially vegan diets, are associated with specific risks and benefits for certain population groups such as pregnant women, breastfeeding mothers and children, COPLANT will also establish appropriate research structures for these groups and include them in the study.

The detailed consumption survey of all study participants is one of the main pillars of the planned study. Of particular importance is the dietary assessment of novel vegan and vegetarian foods, thus an app adapted to the needs of this study was developed. The characterisation of external and internal intakes of nutrients and contaminants within a particular diet will be examined. Large epidemiological projects currently underway in Germany, such as the NAKO Health Study, are unable to answer these questions. In order to prospectively investigate links between diet and the later occurrence of common diseases such as type 2 diabetes, cardiovascular diseases and cancer, the study participants should be followed up for at least 20 years if third-party funding is successfully acquired.

The study is to be conducted in study centers at the Federal Institute for Risk Assessment (BfR), Berlin, the Max Rubner-Institut (MRI) in Karlsruhe, the Rheinische Friedrich-Wilhelms University in Bonn, the Friedrich Schiller University Jena, the Research Institute for Plant-Based Nutrition in Giessen, in cooperation with the Justus Liebig University Giessen and at the universities of Heidelberg, Regensburg and Vienna. Furthermore, the basic examination includes measurements of body composition, bone health, cardiovascular risk factors, diabetes risk, contaminants and lifestyle. Specific aspects of dietary behavior, physical activity and other lifestyle factors will be assessed using questionnaires. For the basic laboratory program, fasting blood, 24-hour urine collection and a stool sample are taken from all study participants.

Participants will be recruited for the baseline study from 2024 to 2027. Follow-up visits are planned at intervals of 5, 10 and 20 years.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 69 years at recruitment (age-stratified recruitment in four age groups (18 to 29, 30 to 39, 40 to 49 and 50 to 69 years) which should be equally distributed across the four diets)
* following their current diet for at least one year
* health insured
* are willing to have blood taken (adults)
* are willing and able to complete questionnaires
* only at Berlin, Jena, Giessen and Karlsruhe sites: pregnant and breastfeeding women were recruited (shortened examination programm)
* only at the Regensburg, Heidelberg, Bonn and Vienna sites: are neither pregnant nor breastfeeding at the time of recruitment
* only at Berlin and Karlsruhe sites: children of adult participants (shortened examination programm without collection of blood, urine, and stool)
* are able to give informed consent to participate in the study
* have given their consent to participate in the COPLANT study

Exclusion Criteria:

* who can no longer be contacted
* who withdraw their consent to participate in the study

Ages: 18 Years to 69 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — We plan to include proportions of women and men (ratio 1:1), whereby a proportion of women of up to 60 % is accepted.
Study Population: Vegans - no consumption of animal products (less than one exception per month)
  Vegetarians
  * no consumption of meat and fish (less than one exception per month)
  * consumption of eggs and/or dairy products (at least once a month)
  Pescetarians
  * no consumption of meat (less than one exception per month)
  * consumption of fish (at least once a month)
  * consumption of eggs or dairy products possible
  Omnivores/ mixed diet - group of non-exposed persons or control group
  - consumption of meat or sausage (at least once a month).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2047-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of diabetes type 2 | 5, 10, 20 years
  Incidence of diabetes type 2

SECONDARY OUTCOMES:
Incidence of cardiovascular diseases | 10, 20 years
  Incidence of cardiovascular diseases
Incidence of cancer | 10, 20 years
  Incidence of cancer
Vitamin B12 | Baseline
  Vitamin B12 (pmol/l)
Holo-transcobalamine | Baseline
  Holo-transcobalamine (pmol/l),
Homocysteine | Baseline
  Homocysteine (µmol/l)
Methylmalonic acid | Baseline
  Methylmalonic acid (µg/l)
Vitamin B1 status | Baseline
  Vitamin B1 (nmol/l)
Vitamin B2 status | Baseline
  Vitamin B2 (µg/l)
Vitamin B6 status | Baseline
  Vitamin B6 (nmol/l)
Vitamin C status | Baseline
  Vitamin C (mg/l)
Vitamin D status | Baseline
  Vitamin D (nmol/l)
Vitamin E status | Baseline
  Vitamin E (µmol/l)
Iron | Baseline
  Iron (µmol/l)
Ferritin | Baseline
  Ferritin (µg/l)
Transferrin | Baseline
  Transferrin (mg/dl)
Zinc status | Baseline
  Zinc (µg/l)
Selenium status | Baseline
  Selenium (µg/l)
Iodine status | Baseline
  Iodine (µg/l)
Blood pressure | Baseline
  Systolic blood pressure (mm Hg), diastolic blood pressure (mm Hg)
Blood lipids | Baseline
  Total cholesterol, LDL, HDL, triacylglycerides (mmol/l)
Fasting insulin | Baseline
  Fasting insulin (mU/l)
Fasting glucose | Baseline
  Fasting glucose (mmol/l)
Glycated hemoglobin (HbA1c) | Baseline
  HbA1c (%)
C-peptide | Baseline
  C-peptide (ng/ml)
Osteocalcin | Baseline
  Osteocalcin (ng/ml)
Ostase | Baseline
  Ostase (µg/l)
Parathormone | Baseline
  Parathormone (ng/l)
N-terminal propeptide of type I procollagen (PINP) | Baseline
  PINP (ng/ml)
C-terminal telopeptide of type I collagen (CTX) | Baseline
  CTX (ng/ml)
Creatinine | Baseline
  Creatinine (mmol/24h)
Uric acid | Baseline
  Uric acid (mg/24h)
Cytstatin C | Baseline
  Cytstatin C (mg/l)
Thyroid stimulating hormone (TSH) | Baseline
  TSH (mU/l)
Free triiodothyronine (fT3) | Baseline
  fT3 (pmol/l)
Free thyroxine (fT4) | Baseline
  fT4 (pmol/l)
Body fat | Baseline
  Body fat (kg)
Skeletal muscle mass | Baseline
  Skeletal muscle mass (kg)
Total Body Water | Baseline
  Total Body Water (l)
Energy intake | Baseline
  Calories per day
Nutrient intake | Baseline
  Milligramm per day
Intake of dietary supplements | Baseline
  Frequencies per day
Intake of medication | Baseline
  Frequencies per day

OTHER OUTCOMES:
Heavy metals | Baseline
  Arsenic, lead, cadmium (µg/l)
Halogenated, polycyclic aromatic hydrocarbons (dioxins) | Baseline
  Dioxins (ng/g lipid)
Mycotoxins | Baseline
  Mycotoxins (ng/ml)
Per- and polyfluoroalkyl substances (PFAS) | Baseline
  PFAS (ng/ml)
Microbiome | Baseline
  16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Ute Nöthlings, Prof, Principal Investigator — University Bonn; Christine Dawczynski, PhD, Principal Investigator — University Jena; Markus Keller, PhD, Principal Investigator — Research Institute for Plant-based Nutrition (IFPE); Michael Leitzmann, Prof, Principal Investigator — University Regensburg; Ina Danquah, Prof, Principal Investigator — University Heidelberg; Maria Wakolbinger, Prof, Principal Investigator — University Vienna; Tilman Kühn, Prof, Principal Investigator — University Vienna; Beate Fischer, PhD, Principal Investigator — University Regensburg; Benedikt Merz, PhD, Principal Investigator — Max Rubner-Institut; Cornelia Weikert, Prof, Principal Investigator — Federal Institut for Risk Assessment
Locations (8):
- University Vienna, Vienna, Austria
- Germany (7):
  - Max Rubner-Institut, Karlsruhe, Baden-Wurttemberg
  - Friedrich-Schiller University, Jena, Thuringia
  - The German Federal Institut for Risk Assessment, Berlin
  - University Bonn, Bonn
  - Research Institute for Plant-Based Nutrition, Gießen, Giessen
  - University Heidelberg, Heidelberg
  - University Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: Undecided
In accordance with the informed consent of the COPLANT participants, pseudonymised study data could be provided to external researchers upon request for cooperation or data-use purposes. In this case, a cooperation or data use agreement must be concluded in advance. The use of COPLANT study data is therefore only possible with a detailed prior justification of its scientific purpose and after agreement of the steering commitee of the COPLANT study.

REFERENCES:
- See also: summary — http://www.bfr.bund.de/de/coplant-studie.html

DOCUMENTS (1):
  • Study Protocol (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT06323538/Prot_000.pdf